CLINICAL TRIAL: NCT06239961
Title: Multi-Component Behavioral Activation, Nutrition, and Activity Intervention for Persons Aging With HIV
Brief Title: Behavioral Activation, Nutrition, and Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ann Gruber-Baldini, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00107100; 5P30AG028747-17 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2024-02-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: Aging; HIV; Social engagement; Nutrition; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The Brief Behavioral Activation (BA) Coaching will involve having lay coaches work with participants remotely (i.e., by phone or videoconference) to identify and schedule values-based, rewarding social engagement and activities and to use strategies to reduce and problem-solve barriers to social connectedness. Participants first review their daily activity patterns, and then chose activity goals, worked on specific implementation plans, and reviewed their successes and areas for improvement. The behavioral activation coach program will be modified to address the needs of people aging with HIV (PAWH) by working with those in the community to tailor the content and mode of delivery. There will be additional modules on physical activity and nutrition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical Activity Coaching (Experimental): The intervention involves physical activity sessions tailored for people with HIV. Participants engage in physical activities targeting health improvement and fall prevention, promoting physical activity self-efficacy and outcome expectations. Coaches identify individual exercise goals, assess access to physical activity options, and focus on safe, unsupervised strength and balance physical activities at home. Tailored exercise materials, including handouts and videos, are accessible through a website. Additionally, participants are encouraged to follow a structured walking program.
  Interventions: Behavioral: Physical Activity Coaching
- Nutritional Assessment (Experimental): Participants will complete a mini nutritional assessment and keep a food diary. Each participant will meet with a registered dietician for an evaluation. The coaching will be personalized based on the dietician's advice and will include information about community resources for food, making sure health options are available, and suggesting diets and recipes for better eating options.
  Interventions: Behavioral: Nutritional Coaching
- Behavioral Activation (Experimental): Participants receive brief BA (Behavioral Activation) coaching through remote interactions (phone or videoconference) with lay coaches. The structured behavioral approach focuses on identifying and scheduling values-based, rewarding social engagements and activities. Coaches assist in overcoming barriers to social connectedness, involving a review of daily activity patterns, setting activity goals, creating implementation plans, and assessing successes and areas for improvement. The program is adapted for individuals aging with HIV, with community collaboration to tailor content and delivery methods.
  Interventions: Behavioral: Social Connection

INTERVENTIONS:
Behavioral: Social Connection — 6 weekly Behavioral Activation Intervention calls with a 1 hour duration for each call.
  Arms: Behavioral Activation
Behavioral: Nutritional Coaching — 4 weekly nutritional coaching calls with a Registered Dietician with a 1 hour duration for each call.
  Arms: Nutritional Assessment
Behavioral: Physical Activity Coaching — 4 weekly physical activity coaching sessions with a 1 hour duration for each call.
  Arms: Physical Activity Coaching

SUMMARY:
This study will explore if a behavioral intervention program to assist people aged 50 and older with HIV is practical. The program includes a coach who talks with participants, encouraging them to be more active, reduce loneliness, and eat healthier.

DETAILED DESCRIPTION:
This study aims to see if a 12-week program called Behavioral Activation (BA) can help people aged 50 and above with HIV by reducing loneliness and boosting social engagement. The program includes physical activity and nutrition guidance and is led by remote coaches. Investigators will recruit participants from the University of Maryland THRIVE program and other HIV centers in Baltimore. Investigators will test the program with 10 people aged 50 and above with HIV to see if it works. If it proves to be helpful and accepted, investigators might move on to a larger study to evaluate it more thoroughly.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of age or older
2. HIV positive diagnosis
3. Montreal Cognitive Assessment score > 13
4. Report minimal level of loneliness, isolation, and/or depression (PHQ9 > 5)
5. Able to consent
6. Ability to read or speak English
7. Attend the UM THRIVE Center or another HIV center in Baltimore

Exclusion Criteria:

1) No severe cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline and Week 16
  Participants will complete the Patient Health Questionnaire - 9 (PHQ-9) at baseline and at the Week 16 follow up visit. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Where total scores of 5 to 9 = mild, 10 to 14 = moderate, 15 to 19 = moderately severe, and 20 = severe depression.
Loneliness | Baseline and Week 16
  Participants will complete the University of California, Los Angeles (UCLA) Loneliness Questionnaire (Version 3) at baseline and at the Week 16 follow up visit. This is a 20-item scale designed to measure one's subjective feelings of loneliness. Participants rate each item on a scale where 1 = Never, 2 = rarely, 3 = sometimes and 4 = Often. Total scores of 20 - 40 are considered low to moderate, 40 - 60 are considered moderate to high, and score above 60 are considered high in terms of loneliness.
Social Isolation | Baseline and Week 16
  Participants will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation Scale at Baseline and at the Week 16 follow up visit, to measure social isolation. Total scores of 0.5 - 1.0 SD (standard deviation) worse than the mean = mild symptoms/impairment, scores of 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment, and scores 2.0 SD or more worse than the mean = severe symptoms/impairment.
Physical Activity (actigraphy) steps | Baseline and Week 16
  Participants will be given a wearable sensor device to track movements. Physical activity will be assessed using number of daily steps walked measured by the wearable sensor.
Physical Activity (actigraphy) sedentary time | Baseline and Week 16
  Participants will be given a wearable sensor device to track movements. Physical inactivity will be assessed using minutes of sedentary time measured by a wearable sensor.
Total Sleep Time (TST) with Actigraphy | Baseline and Week 16
  TST will be measured by a wearable sensor, from baseline to the final week of the intervention.
Sleep Efficiency (SE) with Actigraphy | Baseline and Week 16
  SE will be measured by a wearable sensor, from baseline to the final week of the intervention.
Sleep Onset Latency (SOL) with Actigraphy | Baseline and Week 16
  SOL will be measured by a wearable sensor, from baseline to the final week of the intervention.
Nutritional Intake | Baseline
  Participants will complete the 18-item Mini Nutritional Assessment (MNA®) at the baseline visit. The MNA® is a screening tool to help identify elderly persons who are malnourished or at risk of malnutrition. A score of 12 or greater indicates the person is well nourished and needs no further intervention. A score of 8-11 indicates the person is at risk of malnutrition. A score of 7 or less indicates the person is malnourished.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7 | Baseline and Week 16
  Participants will complete the Generalized Anxiety Disorder scale-7 (GAD-7) at the baseline and week 16 follow up visit. It is a seven-item diagnostic tool, based on the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) criteria, for identifying likely cases of GAD. Where a score of 0 - 4 = minimal anxiety, 5 - 9 = mild anxiety, 10 - 14 = moderate anxiety, and a score greater than 15 = severe anxiety.
Late Life Function and Disability Instrument | Baseline and Week 16
  Participants will complete the Late-Life Function & Disability Instrument (Late-Life FDI). It is designed to assess and be responsive to meaningful change in two distinct outcomes: function and disability.
  Scores approaching 100 signify high levels in ability to perform discrete actions and activities (without assistance), scores approaching 0 signify low levels in ability to perform discrete actions and activities (without assistance).
Engagement in activities | Baseline and Week 16
  Participants will complete the Yale Physical Activity Survey. This survey was developed to determine the type, amount and patterning of physical activity/exercise in older adults. The tool is composed of two sections - (1) amount of physical activity/exercise performed during a typical week in the past month and (2) activities performed in the past month. In section one, participants are handed a checklist of activity categories (work, exercise, and recreational activities) and are asked how often during the past week they performed a particular activity from each category. Higher scores indicate high levels of physical activity, while lower score indicate lower activity levels or more sedentary lifestyle.
Reece 9-item HIV-related Stigma Scale | Baseline and Week 16
  A 9-item instrument with possible scores ranging from 0 (no perceived stigma) to 45 (high perceived stigma). The HIV Stigma Scale was designed to measure the perception of stigma by those who are HIV infected.
Age | Baseline
  Self reported chronological date of birth.
Race | Baseline
  Self reported racial or ethnic background.
Gender at birth | Baseline
  Characterization of male or female based on their biological characteristics when they were born.
Gender identity now | Baseline
  Characterization of male or female based on their self-identified gender.
Sexual preference | Baseline
  Participants self reported sexual orientation.
Education | Baseline
  Self reported completed level of schooling or degree obtained.
CD4 count | Baseline
  A lab measurement of immune function in patients living with HIV.
HIV viral load | Baseline
  Viral load is a marker of response to antiretroviral therapy (ART).
Bone Mineral Density (BMD) | Baseline
  BMD is expressed by the mass of calcium hydroxyapatite present in a given area or volume of bone in a unit of mass/area (g/cm2) or mass/volume (g/cm3), respectively.
  "-2.5 and below" = "Osteoporosis" " -1.1 to -2.5" = "Osteopenia".
Smoking Status | Baseline
  Participants self reported smoking usage.
Blood pressure | Baseline
  Measurement of the force of blood against the arterial walls, to evaluate the impact of interventions on cardiovascular health.
Lipids (Total cholesterol, Low-density lipoprotein (LDL), High-density lipoprotein (HDL), Triglycerides (TG)) | Baseline
  Lipid panel measures all three cholesterol and triglyceride/fat in the blood to assess for CVD risk. >240 mg/dl = High total cholesterol; 130 - 159 md/dl = High LDL; <40 mg/dl = Low HDL; >150 mg/dl = High TG.
Diabetes status | Baseline
  Assessing participants for the presence or absence of diabetes.
Aspirin usage | Baseline
  Assessing whether participants are using aspirin.
Statin usage | Baseline
  Assessing whether participants are using statin medications.
ASCVD Risk Score | Baseline
  10-year risk calculated using the cardiovascular disease risk measures listed to help decide Statin or Aspirin prescription.
Urine Albumin | Baseline
  Urine analysis detects protein and blood in urine, supposed to be filtered by kidney, where Abnormal = "Risk for renal disease"; >30 = "Kidney disease".
Glomerular Filtration Rate | Baseline
  Measures kidney performance based on the amount of blood filtered per minute. Abnormal = "Risk for renal disease"; <60 = "Kidney disease"; <=15 = "Kidney failure".

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gruber-Baldini, PhD, Principal Investigator — UMB
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Because a feasibility study, of 10 persons, the data could be identifiable.